CLINICAL TRIAL: NCT05002413
Title: NANO-RAST: Nanomotion-based Resistell AST to Determine the Antibiotic Susceptibility of Gram-negative Bacteria Causing Bacteremia and/or Sepsis
Brief Title: Nanomotion-based Resistell AST to Determine the Antibiotic Susceptibility of Gram-negative Bacteria Causing Bacteremia and/or Sepsis
Acronym: NANO-RAST
Status: Completed | Type: Observational
Sponsor: Resistell AG (Industry)
Collaborators: Innosuisse - Swiss Innovation Agency (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01622
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Bacteremia Sepsis
Keywords: Bacteremia Sepsis Antibiotic Susceptibility Testing AST Gram-negative; Resistell Phenotech; Nanomotion; Cantilever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Resistell AST — The Resistell AST is intended for rapid antibiotic susceptibility testing of most common clinically relevant Gram-negative bacteria causing bloodstream infections (BSI) (bacteremia). In the scope of this study, the Resistell Phenotech device will be used to test the susceptibility of Gram-negative bacteria, in particular Escherichia coli and Klebsiella pneumoniae to ceftriaxone and ciprofloxacin.
  Other Names: Resistell Antibiotic Susceptibility Test

SUMMARY:
Blood culture samples from bacteremia patients positive for Gram-negative bacteria will be tested for antibacterial susceptibility using Resistell Phenotech device. The results will be compared with current AST gold standard tests to calculate sensitivity, specificity, and accuracy of Resistell Phenotech device.

DETAILED DESCRIPTION:
NANO-RAST: Nano-motion based Resistell AST to determine the antibiotic susceptibility of bacteria causing bacteremia and sepsis.

Study population: patients admitted at the study site with bacteremia considered to be due to a pathogenic strain (E. coli or K. pneumoniae).

Study design: prospective, observational, single arm study.

ELIGIBILITY:
Inclusion Criteria: The patients meeting all the following criteria can be recruited in the study:

* patients over the age of 18 years who sign, or their relatives / legal representatives sign the informed consent form;
* patients with bacteremia considered to be due to a pathogenic strain;
* patients hospitalized at CHUV at the time of blood culture inoculation;
* patients whose positive blood cultures were not older than 24 hours at the time of AST start.

Exclusion Criteria The patients meeting any of the following criteria will be excluded from the study:

* patient is diagnosed with polymicrobial bacteremia;
* samples can be excluded from the study during the processing of samples in case of technical errors e.g. failure with attachment of cells, technical problem with the device or sensor, operator's error, etc.

Note: in the event that the capacity of the Resistell instruments is reached for the day, no more ICFs will be obtained for the day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bacteremia considered to be due to a pathogenic strain who have been hospitalized at CHUV at the time of blood culture inoculation
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Resistell AST | Approximately 30 months
  The primary endpoint will be the sensitivity of the device in detecting antibiotic susceptibility in blood samples positive for Gram-negative bacteria.

SECONDARY OUTCOMES:
Accuracy and Specificity of Resistell AST | Approximately 30 months
  Accuracy and specificity of the device will be calculated to test the effectiveness of the device.
Time to Result (TTR) | Approximately 30 months
  Time to Result (TTR) from the point the blood culture turns positive for Gram-negative bacteria to the point antibiotic susceptibility results are obtained from the Resistell AST device.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de microbiologie CHUV R , Suisse +41 21 314 4056, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caruana G, Kritikos A, Vocat A, Tagini F, Delfino A, Luraschi A, Delarze E, Marta PV, Delaloye J, Jacot D, Winnicki J, Orlando C, Sturm A, Jozwiak G, Cichocka D, Greub G. Nanomotion-based technology for rapid antibiotic susceptibility testing among adult patients admitted to a tertiary-care hospital with Gram-negative bacteraemia: a prospective, single arm, comparative diagnostic accuracy study. Clin Microbiol Infect. 2026 Feb;32(2):299-305. doi: 10.1016/j.cmi.2025.10.016. Epub 2025 Oct 29. PMID 41173335
- [Derived] Caruana G, Kritikos A, Vocat A, Luraschi A, Delarze E, Sturm A, Pla Verge M, Jozwiak G, Kushwaha S, Delaloye J, Cichocka D, Greub G. Investigating nanomotion-based technology (Resistell AST) for rapid antibiotic susceptibility testing among adult patients admitted to a tertiary-care hospital with Gram-negative bacteraemia: protocol for a prospective, observational, cross-sectional, single-arm study. BMJ Open. 2022 Nov 21;12(11):e064016. doi: 10.1136/bmjopen-2022-064016. PMID 36410804